CLINICAL TRIAL: NCT02425735
Title: γδ T Cell Immunotherapy for Treatment of Hepatocellular Liver Cancer
Brief Title: Safety and Efficiency of γδ T Cell Against Hepatocellular Liver Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Jinan University Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Gd T cell and Hepatocellular
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2015-04

CONDITIONS: Liver Cancer
Keywords: Immunotherapy, γδ T Cell, heptocellular liver cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): DC-CIK cells will be used against tumor cells.
  Interventions: Biological: DC-CIK cells
- Group B (Experimental): γδ T cells will be used against tumor cells.
  Interventions: Biological: γδ T cells
- Group C (Experimental): Combination of γδ T cells/ DC-CIK be used against tumor cells.
  Interventions: Biological: γδ T/DC-CIK cells

INTERVENTIONS:
Biological: DC-CIK cells — DC-CIK cells will be used against tumor cells.
  Arms: Group A
Biological: γδ T cells — γδ T cells will be used against breast tumor.
  Arms: Group B
Biological: γδ T/DC-CIK cells — γδ T/DC-CIK cells will be used against breast tumor.
  Arms: Group C

SUMMARY:
In this study, effects of γδT cells on human hepatocellular liver cancer in combination with tumor reducing surgery, for example cryosurgery going to be investigated.

DETAILED DESCRIPTION:
Liver tumor will be removed using tumor reducing surgery such as cryosurgery. PBMC of the patient will be separated from peripheral blood. After making them potential cancer killer γδ T Cell and DC-CIK, they will be infused to the patients as an immunotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-75
2. Karnofsky performance status >50
3. Diagnosis with hepatocellular carcinoma cancer based on histology or the current accepted radiological measures.
4. Classification tumor,nodes,metastasis-classification(TNM) stage: Ⅱ,Ⅲ,Ⅳ
5. Will receive cryosurgery, gd Tcells/ DC-CIK.
6. Life expectancy: Greater than 3 months
7. Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients with other kinds of cancer
2. History of coagulation disorders or anemia
3. Patients with heart disease and diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Reduced size of the tumors | Up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Alnaggar M, Xu Y, Li J, He J, Chen J, Li M, Wu Q, Lin L, Liang Y, Wang X, Li J, Hu Y, Chen Y, Xu K, Wu Y, Yin Z. Allogenic Vgamma9Vdelta2 T cell as new potential immunotherapy drug for solid tumor: a case study for cholangiocarcinoma. J Immunother Cancer. 2019 Feb 8;7(1):36. doi: 10.1186/s40425-019-0501-8. PMID 30736852